CLINICAL TRIAL: NCT02336633
Title: Metabolic Intervention Using Resveratrol in Patients With Huntington Disease
Brief Title: Resveratrol and Huntington Disease
Acronym: REVHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P130918
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-08

CONDITIONS: Huntington Disease
Keywords: Huntington disease; Neurodegenerative disease; Volumetric MRI; 31P MR spectroscopy; metabolism; Caudate atrophy
MeSH Terms: conditions — Huntington Disease; Neurodegenerative Diseases | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Resveratrol (80mg/j = 4 capsules/day)
  Interventions: Dietary Supplement: Resveratrol
- 2 (Placebo Comparator): Placebo (4 capsules/day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — 2 capsules of 20mg in the morning and in the evening (4 capsules in total/day = 80mg/day) every day during 1 year
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the therapeutic potential of Resveratrol on the caudate volume in HD patients, using volumetric MRI.

DETAILED DESCRIPTION:
Thanks to neuroimaging biomarkers already validated in HD and the newly identified metabolic brain biomarkers using 31P-MRS, we can test for a reduction in neurodegeneration among HD patients resulting from an improvement in brain energy profiles with resveratrol.

We plan to randomize 102 early affected HD patients (with a maximum of 120 included patients) in France (5≤UHDRS≤40) in a randomized, double-blind, controlled study. Patients will receive either resveratrol at 80 mg (n=51), or placebo (n=51) for 12 months. Clinical benefit will be respectively evaluated by UHDRS and neuropsychiatric questionnaires; biological tolerance will be evaluated by routine biochemical blood tests and plasma measurements of resveratrol, these three factors will be tested every three months.

The primary end-point will be the measure of the rate of caudate atrophy - the most sensitive biomarker identified to date in HD - after one year of treatment with resveratrol in early affected HD patients using volumetric MRI as we described.

Secondary end-points include:

The clinical and biological tolerance of resveratrol in HD patients will be evaluated by (i) neuropsychiatric questionnaires: Starkstein apathy scale, Hospital Anxiety and Depression Scale (HADS), Systems Behaviour Inventory (FrSBe) and SF36, (ii) a cognitive test; Symbol Digit Modalities Test (SDMT) and (iii) routine biochemical tests The clinical benefit of resveratrol will be evaluated by a decrease in the progression of the UHDRS over a year of treatment The benefit of resveratrol on brain energy metabolism will be evaluated by the restoration of an increased ratio of inorganic phosphate/phosphocreatine - reflecting normal brain activation - during visual stimulation, using 31P-MRS as we described The progression of caudate atrophy over a year will be correlated with the changes in brain energy profile as well as changes in the progression of the UHDRS.

The compliance of treatment and peak in plasmatic concentration through plasma measurements of resveratrol.

ELIGIBILITY:
Inclusion criteria :

* Positive genetic test with CAG repeat length > or = 39 in HTT gene
* At least 18 years of age
* Signature of the informed consent
* Covered by social security
* UHDRS score between 5 and 40 (both included)
* Ability to undergo MRI scanning

Exclusion criteria :

* Hypersensitivity to resveratrol or to one of its excipients (gelatin and glycerin)
* Tetrabenazine treatment
* Neuroleptic treatments other than olanzapine at small doses (≤10 mg) and Abilify® (≤15mg)
* VKA treatment (Previscan®, Sintron®, Coumadine®)
* NACO treatment (Pradaxa®, Xarelto®, Eliquis®)
* Additional psychiatric or neurological conditions
* Severe head injury
* Participation in another therapeutic trial (3 months exclusion period)
* Pregnancy and breastfeeding
* Inability to understand information about the protocol
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-07; Primary Completion 2019-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
rate of caudate atrophy | 1 year
  Measurement of the rate of caudate atrophy before and after one year of treatment with resveratrol in early affected HD patients using volumetric MRI.

SECONDARY OUTCOMES:
UHDRS (Unified Huntington Disease Rating Scale) | 1 year
TFC (Total Functional Capacity) | 1 year
ratio of inorganic phosphate/phosphocreatine | 1 year
  The benefit of resveratrol on brain energy metabolism will be evaluated by the restoration of an increased ratio of inorganic phosphate/phosphocreatine - reflecting normal brain activation - during visual stimulation, using 31P-MRS will be assessed before and after 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Mochel, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut du Cerveau et de la Moelle, Hôpital de la Pitié Salpêtrière, Paris, France